CLINICAL TRIAL: NCT00220571
Title: Combined Abciximab Reteplase Stent Study in Acute Myocardial Infarction
Brief Title: CARESS in Acute Myocardial Infarction
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Società Italiana di Cardiologia Invasiva (Other)
Collaborators: Royal Brompton & Harefield NHS Foundation Trust (Other); Eli Lilly and Company (Industry); Biotronik SE & Co. KG (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IIT(IT) H4S-IT-O038; 2003OE001B
Record Dates: First submitted 2005-09-13; First posted 2005-09-22 (Estimated); Last update posted 2007-07-03 (Estimated); Status verified 2005-09

CONDITIONS: Myocardial Infarction
Keywords: AMI; stent; PTCA; abciximab; reteplase; combo therapy
MeSH Terms: conditions — Myocardial Infarction | interventions — Angioplasty, Balloon

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: Coronary Angioplasty (PTCA)

SUMMARY:
The aim of this study conducted in patients with high risk ST-segment elevation AMI admitted to hospitals with no PTCA facilities is to compare the effects on clinical outcome and cost-effectiveness of two reperfusion strategies:

* Fibrinolytic therapy with Abciximab and half-dose Reteplase, with rescue PTCA in case of lack of reperfusion
* Elective referral for "facilitated" PTCA after early administration of Abciximab and half dose of Reteplase

DETAILED DESCRIPTION:
All patients with ST-segment elevation AMI admitted within 12 hours from symptoms onset will be screened to enter in this study. Data of patients with ST-segment elevation AMI within 12 hours from symptoms onset who do not meet the inclusion criteria or do not sign the informed consent form are entered into a dedicated registry.

ELIGIBILITY:
Inclusion Criteria:

- ECG with ST-elevation (≥ 1mm in at least 2 ECG limb leads or ≥ 2 mm in 2 contiguous precordial leads) AMI within <12 hours from symptoms onset fulfilling 1 or more of the following criteria of "high risk":

1. Summation of ST-segment elevation or depression ≥ 15 mm in all 12 electrocardiographic leads or new onset complete left bundle branch block;
2. Previous myocardial infarction (Q- and non Q-wave);
3. Killip Class 2 or 3;
4. LV ejection fraction at transthoracic ultrasound < 40%.

Exclusion Criteria:

1. Inability to provide informed consent;
2. Age > 75 years
3. CABG or PCI procedure in past history involving the infarct-related artery;
4. Participation in another study with any investigational drug or device within the previous 30 days;
5. Concomitant non-cardiac disease likely to limit long-term prognosis (e.g. cancer);
6. Cardiogenic shock (hypotension with Systolic Blood Pressure (SBP) < 90 mmHg and tachycardia > 100 beats / min, not due to hypovolemia and requiring inotropic support or balloon counterpulsation);
7. Need for concomitant major surgery (e.g. valve surgery or resection of aortic or left ventricular aneurysm, carotid endarterectomy, abdominal aortic aneurysm surgery, congenital heart disease etc);
8. Severe hepatic disease;
9. Patients with acute or chronic renal impairment (serum creatinine > 2.0 mg % or 200 mg/l or creatinine clearance < 30 ml/min);
10. Transmural MI in different location within the previous week;
11. Previous administration of thrombolytics within 7 days;
12. Intolerance or contraindications to ASA or Clopidogrel;
13. Known leucopenia, defined as a leukocyte count of < 3.500 White Blood Cells (WBC)/ml
14. Known neutropenia, defined as < 1000 neutrophils / ml;
15. Known thrombocytopenia (< 100.000 platelets / ml );
16. Documented active peptic ulcer or upper gastrointestinal bleeding within the previous 6 months;
17. Previous hemorrhagic stroke;
18. Previous ischemic cerebrovascular event within 3 months;
19. Intracranial neoplasm;
20. Recent major surgery at risk of bleeding;
21. Episodes of uncontrolled hypertension (> 180/110 mmHg despite treatment) in past 2 years;
22. Administration of oral anticoagulants within the previous 7 days unless INR ≤ 1.2;
23. Severe recent trauma;
24. Known or possible pregnancy;
25. Absence of suitable vascular access (diffuse peripheral arterial disease);
26. Basal ECG changes which make identification of ST-segment elevation impossible (i.e.: ventricular activation from artificial pacemaker, etc.).

Max Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 600 (Actual)
Dates: Start 2003-05; Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
To compare 30 days incidence of the composite end-point of: mortality, reinfarction and refractory ischemia in the two arms of the study. | 30 Day

SECONDARY OUTCOMES:
Compare 1 year composite end-point of: mortality, reinfarction, refractory ischemia, hospital readmission because of heart failure in the two arms; | 1 Year
Compare the resource use at 30 days and 1 year, including days in CCU, MICU or general ward, cost of catheterization and PTCA, drugs, ambulance service during index hospitalization and subsequent hospital admissions for reAMI | 30 Day and 1 Year
Compare the incidence of in-hospital stroke and bleeding complications in the two arms. | 30 Day

CONTACTS AND LOCATIONS:
Overall Officials: Leonardo Bolognese, MD, Ph D, Principal Investigator — Ospedale San Donato - Arezzo Italy; Gabriel P. Steg, MD. Ph D, Principal Investigator — Hopital Bichat - Paris France; Darius Dudek, MD, Ph D, Principal Investigator — Jagellonian University Krakow Poland; Carlo Di Mario, MD, Study Chair — Royal Brompton and Harefield Hospital - London UK
Locations (85):
- France (15):
  - Cardiologie Hop. Duffaut, Avignon
  - SAMU - Hop. Duffaut, Avignon
  - Cardiologie - Hop. Louis Pradel, Bron
  - Cardiologie - CH, Caen
  - Urgences - CH, Carpentras
  - Cardiologie - CH, Cherbourg
  - SAMU - Hop. Beaujon, Clichy
  - Service de Cardiologie - Hopital St. Joseph, Colmar
  - Cardiologie - CHU, Grenoble
  - Samu - Chu, Grenoble
  - SAMU 69 - Hop. E. Herriot, Lyon
  - Cardiologie - Hop. Bichat, Paris
  - Centre Cardiologique du Nord, Saint-Denis
  - SMUR Delafontaine, Saint-Denis
  - SAMU - Reanimation - CH, Sélestat
- Italy (47):
  - Ospedale San Donato, Arezzo
  - Presidio Ospedaliero del Casentino, Bibbiena
  - Spedali Civili, Brescia
  - Az. Ospedaliera di Circolo, Busto Arsizio
  - P.O. di Camposampiero, Camposampiero
  - Ospedale Ramazzini, Carpi
  - Ospedale Bufalini, Cesena
  - P.O. Cittadella, Cittadella
  - P.O. di Codogno, Codogno
  - Ospedale di Conegliano, Conegliano
  - Ospedale S. Giuseppe da Copertino, Copertino
  - Ospedale S. Sebastiano, Correggio
  - P.O. di Cortona, Cortona
  - Ospedale Santa Croce e Carle, Cuneo
  - Ospedale di Desio, Desio
  - Ospedale Santa Maria del Prato, Feltre
  - Ospedale S. Sebastiano Martire, Frascati
  - Ospedale Santa Caterina Novella, Galatina
  - Ospedale La Memoria, Gavardo
  - Ospedale San Giuliano, Giugliano in Campania
  - Ospedale di Guastalla, Guastalla
  - Az. Osp.Vito Fazzi, Lecce
  - Ospedale Civile di Legnano, Legnano
  - Az. Ospedaliera Desenzano sul Garda, Manerbio
  - Fondazione Centro San Raffaele del Monte Tabor IRCCS, Milan
  - Hesperia Hospital, Modena
  - Nuovo Ospedale S. Agostino Estense - Baggiovara, Modena
  - Ospedale Civile, Mondovì
  - P.O. di Montebelluna, Montebelluna
  - Ospedale Franchini, Montecchio
  - Azienda Universitaria Federico II, Napoli
  - Ospedale Santa Maria delle Grazie, Pozzuoli
  - Arcispedale Santa Maria Nuova, Reggio Emilia
  - Ospedale Civile, Riccione
  - Ospedale degli Infermi, Rimini
  - Ospedale S. Eugenio, Roma
  - A.O. San Camillo, Roma
  - Istituto Clinico Humanitas, Rozzano
  - P.O. U.O. Struttura Complessa, San Giovanni Valdarno
  - Ospedale della Valtiberina, Sansepolcro
  - Ospedale Provinciale di Saronno, Saronno
  - Nuovo Ospedale Civile di Sassuolo, Sassuolo
  - Ospedale SS.Annunziata, Savigliano
  - Ospedale M. Scarlato, Scafati
  - Ospedale Magati, Scandiano
  - Az. Ospedaliera Galmarini, Tradate
  - Ospedale Cà Foncello, Treviso
- Poland (23):
  - Specjalista Chorob Wewnetryznich, Będzin
  - Oddzial Chorob Wewnetrznych, Brzesku
  - Szpital Powiatowy w Chrzanowie, Chrzanów
  - Oddzialu Kardiologicznego, Dąbrowa Górnicza
  - Oddzialu Chorob Wewnetrznych, Dąbrowa Tarnowska
  - II Oddzial Kardiologiczno - Wewnetrezny Szpital Miejski w Jawozznie, Jaworzno
  - Oddzial Wewneztrnj Okregowy Szpital Kolciowy, Katowice
  - First Dept. Cardiology - Gornoslaskiego Centrum Medycznego, Katowice
  - Zaklad Hemodynamiki i Angiokardiografii Pracownia 1, Krakow
  - Zaklad Hemodynamiki i Angiokardiografii - Pracownia 2, Krakow
  - Oddzial Wewnetrzny - Szpital Mijski w Krynicy, Krynica
  - Oddzial Wewnetrzny - Szpital Powiatowy w Limanowej, Limanowa
  - Oddzial Internistyczno- kardiologiczny, Nowy Sącz
  - Oddzial Kardiologiczny, Nowy Targ
  - Szpital Powiatowy im. Sw. Maksimiliana w Oswiecimiu, Oświęcim
  - Oddzial Intensywnej Opieki Kardiologicznej i Kardiologii Olgonej, Sosnowiec
  - Zaklad Opieki Zdrowotnej, Sucha Beskidzka
  - Oddzial Wewnetrzny Szpital w Szczyrzu, Szczyrzyc
  - Oddzial Kardiologii Inwazijnej - Szpital im. E. Szczeklika, Tarnów
  - Oddzialu Kardiologii z OIOK, Tarnów
  - Oddzial Kardiologii - Szpital Miejski w Tychach, Tychy
  - Szpital Powiatowy im. Jana Pawla II w Wadowicach, Wadowice
  - Oddzial Kardiologii - Szpital Powiatowy w Zakopane, Zakopane

REFERENCES:
- [Background] Di Mario C, Bolognese L, Maillard L, Dudek D, Gambarati G, Manari A, Guiducci V, Patrizi G, Rusconi LC, Piovaccari G, Hibon AR, Belpomme V, Indolfi C, Olivari Z, Steffenino G, Zmudka K, Airoldi F, Panzarasa R, Flather M, Steg PG. Combined Abciximab REteplase Stent Study in acute myocardial infarction (CARESS in AMI). Am Heart J. 2004 Sep;148(3):378-85. doi: 10.1016/j.ahj.2004.03.038. PMID 15389222
- [Derived] Di Mario C, Dudek D, Piscione F, Mielecki W, Savonitto S, Murena E, Dimopoulos K, Manari A, Gaspardone A, Ochala A, Zmudka K, Bolognese L, Steg PG, Flather M; CARESS-in-AMI (Combined Abciximab RE-teplase Stent Study in Acute Myocardial Infarction) Investigators. Immediate angioplasty versus standard therapy with rescue angioplasty after thrombolysis in the Combined Abciximab REteplase Stent Study in Acute Myocardial Infarction (CARESS-in-AMI): an open, prospective, randomised, multicentre trial. Lancet. 2008 Feb 16;371(9612):559-68. doi: 10.1016/S0140-6736(08)60268-8. PMID 18280326